CLINICAL TRIAL: NCT00625560
Title: Randomized, Open-Labelled Study Evaluating the Antiviral Efficacy, Safety, and Tolerability of Continuing Lamivudine Therapy or Switching to Entecavir in Subjects With Chronic Hepatitis B With Detectable HBV DNA
Brief Title: Continuing Lamivudine vs Switching to Entecavir in Patients With Detectable HBV DNA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0351
Record Dates: First submitted 2008-02-11; First posted 2008-02-28 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; Lamivudine; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): entecavir 1.0 mg QD
  Interventions: Drug: Entecavir
- B (Active Comparator): lamivudine 100 mg QD
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — entecavir 1.0 mg QD
  Other Names: Baraclude 1.0mg
  Arms: A
Drug: Lamivudine — lamivudine 100 mg QD
  Other Names: Zeffix 100mg
  Arms: B

SUMMARY:
This is a randomized, open-labelled, prospective 96-week study comparing the antiviral efficacy and safety of switching to entecavir 1 mg QD from lamivudine versus maintaining lamivudine 100 mg QD treatment in HBV-infected subjects currently receiving lamivudine monotherapy.

DETAILED DESCRIPTION:
Entecavir has a higher potent antiviral efficacy and a lower drug resistance rate than Lamivudine in nucleoside-naïve CHB patients. The prompt switch from Lamivudine to Entecavir in patients who have insufficient hepatitis B virus suppression (HBV DNA ≥ 60 IU/mL by PCR) may lead to full viral suppression to undetectable level by PCR method. The prompt switch from Lamivudine to Entecavir in patients who have insufficient hepatitis B virus suppression (HBV DNA ≥ 60 IU/mL) may preclude development of drug resistance. The results of this study will provide a rationale for switch treatment from one antiviral to another one, especially from LAM to ETV.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-70 years of age) currently taking lamivudine monotherapy for chronic HBV infection for at least 6 months with ≥ HBV DNA 60 IU/mL level and HBeAg positive at baseline.

Exclusion Criteria:

* All subjects will be tested for presence of M204V/I mutations in the YMDD motif at baseline. Subjects with M204V/I mutations in the YMDD motif at baseline are not eligible for the study.
* Subjects treated with other antiviral drugs (e.g. adefovir) in combination with lamivudine are not eligible for this study.
* Subjects should have ALT < 10 x ULN, and no evidence of hepatocellular carcinoma.
* Subjects should be without serological evidence of co-infection with HCV, HIV, or HDV.
* Subjects with decompensated liver disease, as well as pregnant or breast-feeding women, will not be eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage number of patients with HBV DNA < 60 IU/mL (Undetectable serum HBV DNA by PCR method) while on randomized therapy | at Week 96

SECONDARY OUTCOMES:
Percentage number of patients with HBV DNA < 60 IU/mL while on randomized therapy | at Week 48
Percentage number of patients who developed drug resistant mutations while on randomized therapy | at Week 48 and Week 96
Change from baseline in mean HBV DNA | at Week 48 and 96
Percentage number of patients who achieved ALT normalization, HBeAg loss, HBe seroconversion, HBsAg loss and HBs seroconversion | at Week 48 and 96
Cumulative discontinuation rates due to lamivudine or entecavir resistance mutations and clinical breakthrough Safety assessment | Follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, M.D.Ph.D, Study Chair — Yonsei Univsersity College of Medicine; Do Young Kim, M.D., Study Director — Yonsei University; Jun Yong Park, M.D, Principal Investigator — Yonsei University; Jeong Heo, M.D.Ph.D, Study Director — Pusan National University
Locations (2):
- South Korea (2):
  - Pusan National University School of Medicine, Busan, Busan
  - Severance Hospital, Seoul, Seoul